CLINICAL TRIAL: NCT01882153
Title: Evaluating Parent Delivered Interventions for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Associate Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-11232011-8727
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Autistic Disorder; Developmental Disabilities
MeSH Terms: conditions — Autistic Disorder; Developmental Disabilities

ARMS (2):
- Developmentally Based Intervention (Experimental)
  Interventions: Behavioral: PACE Therapy; Behavioral: PACE and PRT Hybrid
- Behaviorally Based Intervention (Experimental)
  Interventions: Behavioral: Pivotal Response Training (PRT); Behavioral: PACE and PRT Hybrid

INTERVENTIONS:
Behavioral: Pivotal Response Training (PRT) — The behaviorally-based intervention is a treatment model that uses the principles of Applied Behavior Analysis (Koegel, Openden, Fredeen, & Koegel, 2006) to increase children's adaptive behaviors and decrease maladaptive behaviors.
  Arms: Behaviorally Based Intervention
Behavioral: PACE Therapy — The developmentally based intervention is grounded in a development theory, that focuses on child-directed interactions with warm and caring individuals that aid in acquiring missed developmental and functional milestones.
  Arms: Developmentally Based Intervention
Behavioral: PACE and PRT Hybrid — The hybrid based treatment has an eclectic approach that incorporates both systematic (behaviorally-based) and affect-based learning (developmentally-based)that focuses on increasing children's skill development (http://www.pacificautism.org).

SUMMARY:
The investigators will assess the efficacy of parent delivered interventions in the treatment of social and communication deficits in children with autism. By collecting information about parent and child functioning before and after intervention, the investigators will be able to determine whether the intervention is effective in improving child social communication and reducing parent stress.

ELIGIBILITY:
Inclusion Criteria for autism participants:

* Children between the ages of 1.6 and 17.11 years of age
* Males and females
* Diagnosis of autism based on DSM-IV-TR criteria, an expert clinical evaluation, and ADOS or ADI-R if needed
* Receiving or will receive a parent delivered intervention to alleviate symptoms related to their diagnosis of autistic disorder
* Have a care provider that will reliably bring subjects to their chosen intervention and clinic visits, and is trustworthy to provide accurate accounts of services provided to the subject

Inclusion Criteria for developmentally delayed participants:

* Will have an age range between 1.6 and 17.11 years of age
* Males or females
* Diagnosis of a developmental delay or disorder based on DSM-IV-TR, ICD-10, and an expert clinical evaluation
* Have historical evidence of significant abnormal developmental milestones as determined by neurological history
* Receiving or will receive a parent delivered intervention
* Have a care provider that will reliably bring subjects to their chosen intervention and clinic visits, and is trustworthy to provide accurate accounts of services provided to the subject

Exclusion Criteria for autism participants:

* Is medically unstable (e.g., more than one seizure a month)
* Have a medical diagnosis that causes autism like symptomology (e.g., Fragile X, Down syndrome, Angelman's syndrome, tuberous sclerosis, Rett's disorder)

Exclusion Criteria for developmentally delayed subjects:

* Is medically unstable (e.g., more than one seizure a month)
* Has a diagnosis of ASD

Ages: 18 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Change in CGI-S (Clinical Global Impression - Severity) | Difference from Baseline to Week 12
Change in SRS (Social Responsiveness Scale) | Difference from Baseline to Week 12
Change in CDI (Communicative Development Survey) Score | Difference from Baseline to Week 12
Change in social and communication behaviors as assessed by standardized laboratory observations | Difference from Baseline to Week 12

SECONDARY OUTCOMES:
Change in VABS (Vineland Adaptive Behavior Scale) Score | Difference from Baseline to Week 12
Change in social and communication behaviors as assessed from home videos | Difference from Baseline to Week 12
Change in PSI (Parenting Stress Index) Score | Difference from Baseline to Week 12
Change in FES (Family Empowerment Scale) Score | Difference from Baseline to Week 12
Change in frequency and duration of investigation therapy | Difference from Baseline to Week 12
Change in demographics data | Difference from Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y Hardan, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States